CLINICAL TRIAL: NCT02538406
Title: The Utility of Time Segmental Withdrawal During Screening Colonoscopy for Increasing Adenoma Detection Rate. A Randomized Controlled Clinical Trial.
Brief Title: The Utility of Time Segmental Withdrawal During Screening Colonoscopy for Increasing Adenoma Detection Rate.
Status: Terminated | Type: Observational
Why Stopped: Local IRB in process to close down study.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, M.D. Director of Advanced Endoscopy Assistant Professor of Medicine - Gastroenterology Section, Baylor College of Medicine
Other Study IDs: H-37320
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Adenomatous Polyp of Colon
Keywords: Adenoma; withdrawal time; Colonoscopy
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non segmental withdrawal: A standard of care colonoscopy will be done on the patient without extra time on the right side of the colon.
- Segmental withdrawal: A standard of care colonoscopy will be done on the patient , however the time spent in the right side of the colon will be more than half of the normal colonoscopy procedure (i.e. more than 3 minutes)
  Interventions: Other: Segmental withdrawal

INTERVENTIONS:
Other: Segmental withdrawal — Interventional group will have at least 3 minutes dedicated to the right side of the colon during segmental withdrawal.
  Groups: Segmental withdrawal

SUMMARY:
Colonoscopy( examining the colon with a flexible tube and a camera ) is usually done for screening purposes to find any precancerous lesions (polyps) at an early stage. During the colonoscopy the doctor will advance the colonoscope to the end of your colon and start examining the colon for any polyps. "Withdrawal time" is the period of time the doctor spends examining the colon. Doctors usually spend six minutes examining the colon after they reach the end of the colon. Studies have showed that spending more withdrawal time detects more lesions. The proposal to dedicating half of the withdrawal time during colonoscopy in examining the right side will increase the detection of polyps in the right side of the colon. There will be no other changes in the procedural aspect of the colonoscopy.

DETAILED DESCRIPTION:
Screening colonoscopy is an essential diagnostic tool in the early detection of precancerous colonic lesions, preventing the progression of these lesions to cancer. Population-based and case control studies found a 50% reduction in colo-rectal cancer (CRC) incidence and up to a one-third reduction in mortality from CRC after screening colonoscopy. The effectiveness of colonoscopy in preventing colon cancer is dependent on the adenoma detection rate (ADR) during the procedure. Studies have demonstrated that withdrawal times of 6 minutes or more had higher rates of detection of any neoplasia. In 2006 joint task force of the American College of Gastroenterology and American Society for Gastrointestinal Endoscopy changed the recommendation to indicate that average withdrawal time should exceed 6 minutes in normal colonoscopies in which no polypectomies or biopsies were performed. Based on this recommendation, the 6-minute benchmark is the current standard of care. Longer mean withdrawal times are associated with increasing adenoma detection, mainly of small or right-sided adenomas and proximal serrated adenomas, presumably due to longer inspection of the right colon. However, it also have been showed withdrawal time using 6 minutes as the threshold is not a strong predictor of the likelihood of finding a polyp during colonoscopy and should not be used as a quality indicator. New CRC diagnosis within 3 years of negative screening colonoscopy can be as high as 6%. Right-sided lesions, flat polyps, and variability in endoscopist quality measures are all potential reasons why interval cancers develop. A recent observational study was published showing increase in ADR after implementation of a protocol of careful inspection during a minimum of 8 minutes was established. The investigators hypothesized that if colonoscopists would spend at least half of the time of the withdrawal time in the right side of the colon (referred as segmented protocol), ADR can increase mainly due to the detection of lesions in the right side, which could have been missed otherwise. The investigators are conducting a single center randomized trial investigating the utility of timed segmental withdrawal of at least 3 minutes each in both right and left side of the colon respectively, compared to the regular 6 minutes total withdrawal time regardless of where the time was spent in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-80 years) who are undergoing colonoscopy for screening or surveillance purposes.

Exclusion Criteria:

1. Patients with a prior history of colonic surgeries
2. Patient with Crohns colitis or ulcerative colitis
3. Patient with prior history of colon cancer
4. Patient with poor bowel preparation
5. Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from patients ages 18-80 scheduled for a screening colonoscopy at Baylor College of Medicine. Informed consent will be obtained from the patients during their Gastroenterology clinic visit if the procedure scheduled by gastroenterologist or during their pre-procedure assessment appointment if they were referred by a primary care doctor. Participation in the study will be voluntary. We use the split prep protocol in preparation for colonoscopy in all patients undergoing colonoscopy in our unit.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-08; Primary Completion 2020-06 (Estimated); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Increase in detection rate of adenomas in the right side of the colon | 30 minutes
  To determine if timed segmental withdrawal protocol can increase the adenoma detection rate in the right side of the colon compared to non segmental withdrawal.

SECONDARY OUTCOMES:
Sessile Serrated lesion detection rate | 30 minutes
  Compare sessile serrated lesion detection rate between patients undergoing a screening colonoscopy with segmental withdrawal protocol and non-segmental withdrawal protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O. Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States